CLINICAL TRIAL: NCT06808048
Title: Neurobehavioral Impacts of Medical Cannabis Use: An Observational Study
Brief Title: Medical Cannabis and Behavior
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00011239; R01DA059961 (NIH)
Record Dates: First submitted 2025-01-14; First posted 2025-02-05 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain Patients; Medical Cannabis Users
Keywords: cannabis; medical cannabis; brain MRI; pharmacokinetics
MeSH Terms: conditions — Marijuana Abuse | interventions — Neuropsychological Tests

STUDY DESIGN:
Intervention Model Description: This study is classified by NIH as a basic experimental study of humans (BESH) clinical trial. Enrolled participants are chronic pain patients, some of whom have been prescribed medical cannabis. The study team is not involved in the prescribing of medical cannabis. The interventions to be used in the study are laboratory-based cognitive tests as well as cognitive tasks administered while functional brain activity is recorded. All participants will be administered these measures at a baseline assessment and again after four months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental cognitive and fMRI-based tasks (Experimental): One primary aim of this study is to examine cognitive functioning in individuals who use medical cannabis. All participants in the study will complete cognitive measures that include measures of attention, learning, memory and executive function. All participants will complete task fMRI-based measures of learning and inhibitory control. NIH considers the cognitive and fMRI tasks to be interventions. The fMRI learning task measures face-name associative learning. The fMRI inhibitory control task is a go/no-go task whereby participants respond on some trials to "go" stimuli and withhold responses on other trials to "no-go" stimuli. Brain activations are measured in response to each task. Each participant will complete two cognitive testing sessions as well as two fMRI sessions during the course of the study.
  Interventions: Behavioral: Cognitive testing; Behavioral: Task-based fMRI measure of inhibitory control; Behavioral: Task-based fMRI measure of face-name learning

INTERVENTIONS:
Behavioral: Cognitive testing — Participants will complete a cognitive testing battery that includes measures of attention, learning, memory, problem-solving and executive function.
Behavioral: Task-based fMRI measure of inhibitory control — All participants will complete a task-based fMRI measure of inhibitory control. This Go/No-Go task provides a contrast of BOLD signals when response conflict is low (execution of motor responses on frequent Go trials) vs high (inhibiting the prepotent response on infrequent NoGo trials). It will provide an assessment of the effects of cannabis use on the frontostriatal implicit motor learning and cognitive control systems. Participants view shapes and press a button quickly (Go trials) to every shape except circles and squares (NoGo Trials). To increase response prepotency, Go trials are frequent (75%). Button presses must be rapid to be considered correct. The task uses an event-related design with each stimulus presented for 600 ms, followed by a 1.0-4.5 second jittered ISI during which a white fixation crosshair is displayed. Trial type is pseudo-randomized with the constraint of equal frequencies of consecutive Go trials (2, 3, or 4) between NoGo trials.
Behavioral: Task-based fMRI measure of face-name learning — This task is ideally suited to assess cannabis effects on explicit associative learning and memory as mediated by frontohippocampal networks. Participants memorize names corresponding to faces (encoding phase), and then recall the names after a short delay. The first encoding block begins with a 2-second cue ("MEMORIZE") followed by 5 face-name pairs, each shown for 4 seconds; participants press a button when they encode each face-name pair. A distractor block follows. Next, a retrieval block begins with a cue to "RECALL" followed by presentations of each of the same 5 faces, now paired with "???" (i.e., prompting recall of previously paired names), with a 4 second stimulus duration and no ISI. On recall trials, participants press a button to indicate that they have recalled the name for the displayed face. Participants engage in silent uncued recall of face-name pairs. Immediately following the scan, participants are tested for accuracy of name retrieval.

SUMMARY:
This study will assess cognition, neural function, and drug exposure in chronic pain patients who have been prescribed medical cannabis and will differentiate outcomes based on use of specific CBD-dominant versus THC-dominant treatment products. This longitudinal study will recruit medical cannabis users from local dispensaries. Each participant will complete a baseline assessment prior to the start of medical cannabis use, monthly phone calls to assess treatment adherence, and a four-month follow- up assessment. The aims of this project are: Aim 1. To assess impacts of medical cannabis compounds on executive functions, learning and memory in adults to determine whether cognitive impairments are evident after the onset of cannabis use; Aim 2. To assess the impacts of medical cannabis compounds on white matter microstructure, functional brain activity and functional connectivity; Aim 3. To differentiate change over four months in these outcomes as a function of (a) age and (b) pre-to-post-treatment changes in blood levels of cannabinoid compounds.

DETAILED DESCRIPTION:
This project was submitted to NIH in response to NOT-DA-22-003, Public Health Research on Cannabis. The overarching aim is to assess cognition, neural function, and SUD risk in a sample of patients treated with medical cannabis products in Minnesota (n=120) as compared to non-cannabis using controls (n=60) and to differentiate outcomes based on prescribed doses and blood concentrations of THC versus CBD as objective measures of drug exposure. Patients will be aged 35-65 and qualified for medicinal cannabis treatment in Minnesota due to diagnoses of chronic pain. While deficits in learning, memory and executive functions are reliably observed in young adult recreational cannabis users, it is unclear whether similar impairments characterize individuals who use cannabis for medical reasons, whether adults may be uniquely vulnerable to cannabis-related impairments or if, in fact, use in this age group might be neuroprotective. There are very few published studies of medical cannabis users that comprehensively focus on neurobehavioral outcomes even though at least 5 million people are registered for medical cannabis treatment in the United States. The current study will address this gap through a pre-post assessment of users as compared to matched controls (pain patients who do not use cannabis). Participants will be recruited through posted advertisements and through dispensaries via a collaboration with a local supplier of medical cannabis. They will complete a comprehensive pre-treatment behavioral assessment as well as multimodal brain MRI assessments. All measures will be repeated after four months of treatment. Participants will be interviewed monthly by phone in the interval between visits to assess treatment adherence, pain levels, quality of life, and substance use. Blood cannabinoid levels will be measured at baseline and after four months and will be correlated with behavioral and neural outcomes. The three aims are (1) To assess impacts of medical cannabis compounds on cognition and behavior in otherwise cannabis-naive adults to determine whether impairments that characterize younger users are evident after the onset of medical cannabis use; the investigation will also measure treatment-related changes in pain using well-validated measures. (2) To similarly assess the impacts of medical cannabis compounds on white matter microstructure, functional brain activity and functional connectivity using diffusion-weighted scans, task-based fMRI, and measures of resting state connectivity; (3) To differential change over time in these outcomes as a function of (a) exposure to distinct cannabinoids (THC vs. CBD) as assessed through blood concentrations and (b) age. Sex as a biological variable will be assessed as a covariate of interest. Thus, this proposal will yield a rich dataset through which medical cannabis effects on adults' neurobehavioral function can be assessed and contrasted with the literature on non-medical users.

ELIGIBILITY:
Inclusion Criteria:

* Medical cannabis users (n=120) will be required to

  1. Be ages 35-65;
  2. Be qualified for a medical cannabis prescription based only on a diagnosis of chronic pain; note that individuals can, in theory, utilize medical cannabis for more than one qualifying condition. People with orthopedic pain will be prioritized.
  3. Have normal or corrected-to-normal vision and hearing;
  4. Be free of current and past DSM-V-deﬁned substance use disorders; have < 5 lifetime recreational uses of illicit drugs.
  5. Have limited daily exposure to nicotine (e.g., no daily smokers/vapers; use of nicotine products fewer than 5 occasions weekly);
  6. Willing to abstain from alcohol, nicotine, and other (non-treatment) drugs for 24 hours prior to study. Abstinence will be verified by breathalyzer and urine drug screening; must not test positive on breathalyzer and urine drug screenings for any nonprescribed psychoactive substance or for cannabis (at baseline);
  7. Must be right handed as assessed by the Edinburgh Handedness Inventory;
  8. Lifetime use of cannabis < 15 times; no cannabis product use (recreational or therapeutic) within the past six months;
  9. Able to schedule and complete a multi-hour single session protocol;
  10. Have sufficient manual mobility to be able to complete computerized neurocognitive assessments;
  11. Able to communicate with the researchers by phone during the four month pre-post assessment interval

Pain patients who are not using medical cannabis (n=60) will be required to:

1. Be ages 35-65;
2. Suffer from a chronic pain condition that could qualify them for medical cannabis; People with orthopedic pain will be prioritized.
3. Have normal or corrected-to-normal vision and hearing;
4. Be free of current and past DSM-V-deﬁned substance use disorders; have < 5 lifetime recreational uses of illicit drugs.
5. Have limited daily exposure to nicotine (e.g., no daily smokers/vapers; use of nicotine products fewer than 5 occasions weekly);
6. Willing to abstain from alcohol, nicotine, and other (non-treatment) drugs for 24 hours prior to study. Abstinence will be veriﬁed by breathalyzer and urine drug screening; must not test positive on breathalyzer and urine drug screenings for any non- prescribed psychoactive substance or for cannabis (at baseline);
7. Must be right handed as assessed by the Edinburgh Handedness Inventory;
8. Lifetime use of cannabis < 15 times; no cannabis product use (recreational or therapeutic) within the past six months;
9. Able to schedule and complete a multi-hour single session protocol;
10. Have suﬃcient manual mobility to be able to complete computerized neurocognitive assessments;
11. Able to communicate with the researchers by phone during the four month pre-post assessment interval Within both groups, concomitant opioid use will be allowed as will other prescribed treatments. Controls will be matched to the cannabis group on age, sex, socioeconomic status (SES), type of pain condition (orthopedic pain will be targeted) and comorbid opioid use.

All potential participants must indicate at the baseline enrollment that they have no immediate plans to relocate from the Twin Cities metro area (e.g., must be willing and able to participate in longitudinal assessment for a four-month period).

Exclusion Criteria:

1. Cannot have a degenerative neurological condition or a neurological condition that impacts brain function (e.g., epilepsy);
2. No contraindications to MRI scanning;
3. No lifetime history of severe DSM-V psychopathology (psychotic disorders, bipolar disorder); if currently treated mood for anxiety disorders, must be stable;
4. No current pregnancy or pregnancy within the prior 3 months; cannot be lactating;
5. No cannabis product use (recreational or therapeutic) within the past six months;

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2029-07-15 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Rey Auditory Verbal Learning Test | Administered at baseline and after four months
  All participants will complete a cognitive task battery measuring processes such as learning and memory. The Rey Auditory Verbal Learning Test requires individuals to learn a list of words across five learning trials followed by a distractor list then immediate recall of the initial word list then a 30-minute delayed recall. The minimum score on each trial is 0 and the maximum score on each trial is 15. Scores are tabulated for each of the eight trials. Scores on trials 1-5 reflect learning. Scores on trials 7 and 8 reflect immediate and delayed recall.
Digit Span Task | Administered at baseline and after four months
  The digit span task is a measure of working memory and has a forward and a backward condition. On the forward condition, participants are presented with sequences of digits that are read aloud, beginning with two digits, which the participant must repeat in order. The sequence increases by one digit for each correct level of performance up to a maximum of 9 digits. On the backward condition, the presentation of digits is the same but participants must recall the digit sequences in backward order. The maximum forward and backward span that was correctly recalled is tabulated (min = 0; max = 9).
Verbal Fluency Task | Administered at baseline and after four months
  Participants are told that they will hear a letter (e.g. F) and must generate as many words as they can that begin with that letter in a one-minute period while adhering to certain task rules. Three letters are presented in total, and the total number of words generated without errors is recorded for each letter (min = 0; max = unspecified).
Spatial Span Task | Administered at baseline and after four months
  The spatial span task is a measure of working memory for locations and has a forward and a backward condition. On the forward condition, participants are presented with sequences of targeted locations, beginning with two, which the participant must repeat in order by touching those locations on a computer screen. The sequence increases by one location for each correct level of performance up to a maximum of 9 locations. On the backward condition, the presentation of locations is the same but participants must recall the spatial sequences in backward order. The maximum forward and backward spatial span that was correctly recalled is tabulated (min = 0; max = 9).
Grooved Pegboard Task | Administered at baseline and after four months
  This task is a measure of fine motor coordination. Participants are provided with a board upon which 25 small holes are inserted. They are provided with small pegs to be inserted into the holes. They must place pegs one-by-one into the holes using first the dominant hand and then the non-dominant hand. Dropped pegs are recorded as errors (0 to 25). Completion time (in seconds; min = unspecified; max = 300) is recorded for each hand and is the primary metric that is examined to assess fine motor function and the presence of lateralized motor difficulties.
CANTAB Spatial Paired Associates Learning Task | Administered at baseline and after four months
  Participants view a computer screen on which some number of boxes is displayed in a circular pattern. Boxes are "opened" in a randomized order, one by one. One or more of them will contain a pattern. Participants must learn which patterns go in which boxes. After all box-pattern pairs are shown, the patterns are then displayed in the middle of the screen, one at a time and the participant must select the box in which the pattern was originally located. If the participant makes an error, the boxes are opened in sequence again to remind the participant of the locations of the patterns. Increased difficulty levels (arrays with a greater number of boxes) can be used. Specifically, participants complete up to 5 stages, which involve learning one, two, three, six or eight pattern-location pairings. Outcome measures include the errors made by the participant (max score is unspecified), the number of trials required to locate the pattern(s) correctly, and the number of stages completed.
CANTAB Stockings of Cambridge Task | Administered at baseline and after four months
  This task is a computerized measure of planning ability. On each trial, the participant is shown two displays. In each of these displays, three columns - each containing three colored balls - are suspended from a beam. The two displays appear at the top and bottom of the screen. The balls are arranged in different patterns in each display.The participant must move the balls in the bottom display to match the pattern shown in the top display. The balls are moved one at a time by selecting the required ball, then selecting the position to which it should be moved. The participant is instructed to make as few moves as possible to match the two patterns and is told how many moves are optimal.
  Trials increase in difficulty from 2-move to 5-move problems. Outcomes include the number of problems perfectly solved (max = 12), the number of moves used to execute each problem, and planning time (in milliseconds; how much time the participant waited before beginning to execute each problem).
CANTAB Self-Ordered Search Task | Assessed at baseline and after four months
  On each trial of this working memory task, participants view an array of boxes on a computer screen. Participants search for tokens hidden inside of the boxes. Touching a box reveals whether a token is present. The array size varies from 2 to 8 boxes. When a token is found, it is placed at the side of the screen, and participants are instructed not to return to a location that was previously targeted. Returning to a previously targeted location is a forgetting error. Thus, they must remember where they have searched and found tokens on each trial. For each difficulty level (trials of 3, 4, 6 and 8 boxes), the number of forgetting errors is recorded (high scores = more error). Across 6 and 8-item searches, a strategy score is computed to reflect the extent to which the participant used an organized search strategy. High scores reflect decreased strategy use. Both scores are normed, yielding age-scaled percentiles. CANTAB documentation does not provide max values for the raw scores.
Iowa Gambling Task (IGT) | Assessed at baseline and after four months
  The IGT measures reward-related decision-making. On each of 100 trials, participants select from one of four cards presented on a computer screen. After the selection, feedback is provided. Participants are told that they have won points and, possibly, that they have lost points. Over the course of 100 trials, participants must use this feedback to determine which of the four decks are advantageous (yielding net gains) or disadvantageous (yielding net losses). There are two of each. Outcome measures include the total number of advantageous minus disadvantageous choices across all 100 trials (min = 0; max = 100) as well as for each of five blocks of 20 trials (min score on each block = 0; max = 20). High scores indicate better performance, and the slope of scores across the five blocks indicates rate of learning. Scores will be examined as a function of cannabis use.
Face-Name Learning Task. | Administered at baseline and after four months
  The Face-Name Learning Task will be administered while neural activity is measured. During the task, participants will be presented with ten faces, each of which will be paired with a name. They are asked to memorize the face-name pairings. After all 10 pairs are presented, there is a short delay after which each face is presented alone without the name. Participants are asked to silently recall the name that was associated with the face. Neural activation throughout the brain is measured during the encoding (memorization) phase as well as the recall phase to determine which neural networks are active during these cognitive processes. Activation patterns are then analyzed and contrasted between individuals.
Go No-Go Task of Inhibitory Control | Administered at baseline and after four months
  This task will be administered while neural activation is recorded. During each trial of the task, participants view shapes and press a button quickly (Go trials) to every shape except circles and squares (NoGo Trials). NoGo trials require inhibitory control, because the participant must inhibit the urge to make a response. To increase response prepotency, Go trials are frequent (75%). The task uses an event-related design with each stimulus presented for 600 ms, followed by a 1.0-4.5 second jittered ISI during which a white fixation crosshair is displayed. Trial type is pseudo-randomized with the constraint of equal frequencies of consecutive Go trials (2, 3, or 4) between NoGo trials. This reduces No-Go stimulus predictability and permits an analysis of how increases in response prepotency (longer strings of Go stimuli) impact commission errors (responses to No-Go stimuli). Response accuracy and brainwide neural activity is recorded on each trial.
Intrinsic functional brain activity | Administered at baseline and after four months
  Participants will complete a resting state MRI scan to yield brainwide measures of neural activity at rest. These neural signals form patterns that can be analyzed to differentiate patterns of activation within and between distinct functional networks. These activations will be associated with other behaviors measured in the study, including cannabis use. For this project, activations within the brain's executive control, salience, and reward networks are of maximal interest and will be quantified
MRI measurement of cortical thickness and white matter volume | Administered at baseline and after four months
  Participants will complete structural MRI scans to yield measures of neural structure (gray and white matter volumes and cortical thickness). Images will be acquired for the entire brain and processed to yield cortical thickness (mm), gray matter (volume mm) and white matter (volume mm) for 138 cortical parcels (regions) and 40 subcortical regions.
Frontostriatal structural and functional neural connectivity | Assessed at baseline and after four months
  To assess frontostriatal structure and function, FreeSurfer's segmentation of striatal nuclei (dorsal striatum/caudate; ventral striatum/nucleus accumbens) will be registered to EPI scans to generate seed regions for analyses of frontostriatal structural (diffusion) and functional (fMRI) connectivity. Connections between the dorsal and ventral striatum and discrete regions of the frontal cortex will be quantified and analyzed in relation to performance on the Go No-Go inhibitory control task and as a function of cannabis use over time.
Frontohippocampal structural and functional connectivity | Assessed at baseline and after four months
  Brain MRI T1 and T2 scans will be processed using FreeSurfer, yielding brain-wide cortical parcellations (available across several standard atlases) and subcortical segmentation, which in turn can be employed as ROIs for quantification of diffusion and functional scans following structural-to-EPI registrations. To assess hippocampal structure and function, FreeSurfer's segmentation of hippocampal subfields (based on the high- resolution T2-weighted hippocampal anatomical scan) will be registered to EPI scans to generate seed regions for analyses of frontohippocampal structural (diffusion) and functional (fMRI) connectivity. Anterior-to-posterior (head to tail) hippocampal gradients in structural and functional connectivity will be analyzed with regard to performance on tests of verbal and Face-Name learning as a function of cannabis exposure.
Cannabis Use Disorder Identification Test (CUDIT) | Baseline and monthly for four months thereafter
  Participants will complete an 8-item questionnaire that asked about problems associated with their use of medical cannabis. Each question is rated on a five-point scale (0-4) where high scores indicate increasing frequencies of use or more problematic patterns of use. Scores are summed across the 8 questions to yield a total score, ranging from 0 to 40. Scores of 8 or more indicate hazardous cannabis use, while scores of 12 or more indicate a possible cannabis use disorder.
Blood levels of cannabinoid compounds | Collected at baseline and after four months
  Participants will provide blood samples at the study baseline and four months post-baseline for the measurement of blood cannabinoid levels.
Structured Clinical Interview for DSM-V Substance Use Module | Assessed at baseline and after four months
  The SCID-V Substance Use Module is a semi-structured interview that queries the use of substances of abuse (alcohol, cannabis, stimulants, sedatives, opioids, hypnotics) and the extent to which 11 symptoms of substance use disorder, as defined by the Diagnostic and Statistical Manual of Mental Disorders V, are present for each substance currently and in the past. For each substance, answers to the 11 symptom questions are scored on a three-point scale (0 = absent; 2 = present at subthreshhold level; 3 = present). The full endorsement of two or more symptoms (scores of 3) for each substance class indicates the presence of a substance use disorder (SUD). Three outcome measures that will be analyzed include (1) presence/absence of a SUD for each class of substance, (2) total symptom scores (number of symptoms positively endorsed with ratings of 3) and (3) total symptom scores (summed scores on the 1-3 scale across 11 items for each substance class; min score = 11; max score = 33).
Daily Medication Diary | Daily for the four month duration of the study
  Participants will complete daily diaries across a four-month period to indicate prescription and non-prescription medications that they are ingesting and in what doses. Average daily doses of each medication type, including medical cannabis products, will be quantified and used as outcome measures in data analyses. Minimum possible values = 0; maximum = unspecified.

SECONDARY OUTCOMES:
Alcohol Use Disorders Identification Test (AUDIT) | Baseline and monthly for four months thereafter
  Participant alcohol use will be measured over time using the AUDIT, a 10-item screening tool developed by the World Health Organization (WHO) to assess alcohol consumption, drinking behaviors, and alcohol-related problems. Participants rate each item on a five point scale (0 to 4), and scores are summed across all 10 items to yield an index of problematic alcohol use (min score = 0; max score = 40). A score of 8 or more is considered to indicate hazardous or harmful alcohol use.
Brief Pain Inventory | Baseline and monthly for four months thereafter
  Participants will complete the Brief Pain Inventory to assess their current pain levels and pain-related quality of life. This self report questionnaire asks patients to rate (a) four pain items (worst pain in 24 hours; average pain; least pain in 24 hours; pain right now) and (b) Extent to which pain interferes with general activity, mood, walking ability, sleep, normal work, relations with other people, and enjoyment of life. Each item is rated on a 10-point scale with 1 reflecting low/less pain scores and 10 reflecting high/high pain/high interference with life scores. In addition to scores on individual items, three scores are derived, one that sums responses to the four pain items (max score = 40) and one that sums responses to the interference items (max score = 70) and a total score (sum of all items; max score = 120). High scores reflect worse pain-related impairment.
Beck Depression Inventory (BDI) | Assessed at baseline and monthly for four months
  The BDI is a 21-item self report questionnaire that assesses symptoms of clinical depression and their severity, each rated on a four point scale (0 = symptom is absent; 3 = full presence of the symptom). The questions assess mood and motivation, cognitive symptoms, suicidality, and vegetative symptoms (sleep; libido; eating/weight). Scores are summed across all 21 items to yield a depression severity score (range from 0 to 63). Scores above 21 indicate moderate to severe depression.
UPPS-P Impulsive Behavior Scale | Assessed at baseline and after four months
  The UPPS-P is a 59-item self-report questionnaire that measures five facets of impulsivity (sensation seeking (12 items; scores range from 12 to 48); positive urgency (14 items; scores range from 14 to 56 ); negative urgency (12 items; scores range from 12 to 48); lack of premeditation (11 items; scores range from 11 to 44); lack of perseverance (10 items; scores range from 10 to 40)). Each question is endorsed on a four point scale (1 = strongly agree; 4 = strongly disagree), and the five metrics are derived after implementing reverse-scoring on some items. These five facets of impulsivity will be examined before versus after use of medical cannabis.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Per NIH regulations, data from this project will be shared in a repository. The following types of data will be collected from 180 research participants (chronic pain sufferers who do and do not use medical cannabis): demographic information, lab measures of cognitive performance, self-reported health history and medication use, substance use assessments, multimodal MRI assessments, and biological specimens for the quantification of blood cannabinoid concentrations. Each participant will complete two study visits, during which these measures will be collected, and three interim monthly phone calls during which data on medication use, affect, sleep and pain will be collected. Participants will consent to sharing of their de-identified data. Data will be de- identified prior to receipt by the repository. This study's de-identified data will be shared within the Open Science Framework (OSF), an open platform that facilitates resource sharing and collaboration among registered users.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be curated in an ongoing manner once data collection has been initiated and deposited to the OSF at the conclusion of the performance period and sooner in the context of each publication. The OSF will make decisions about how long to preserve the data. Data made public on OSF is supported by the COS preservation policy: COS established a $400,000 preservation fund for hosted data in the event that COS had to close. If activated, the preservation fund will preserve and maintain read access to hosted public data. This fund is sufficient for many years of read access hosting at present costs beyond the current COS hosting. COS will incorporate growth of the preservation fund as part of its funding model as data storage scales. The dataset generated by this project uses the Open Science Framework (OSF), a free research collaboration/management platform that can be accessed via the OSF API at the address below. The OSF and OSF API are open-source software.
Access Criteria: The data generated by the project will be made available through the OSF JSON API, using the JSON API v1 specification (https://jsonapi.org/format/1.0/). OSF utilizes a unique metadata model that facilitates FAIRness (Findable, Accessible, Interoperable, Reusable) as well as enabling connections across the research lifecycle. The OSF Metadata Profile describes the community vocabularies and persistent identifiers that the OSF uses, the relationships available between metadata fields, the metatags used to enable enhanced web discovery, and an overall map of the metadata implementation. The metadata for the OSF data uses many common metadata standards, and the metadata profile for OSF data can be found at https://help.osf.io/article/573-osf-metadata-profile. There are no substantial limitations on the extent to which this project's data can be shared. Raw neuroimaging files will not be shared. OSF requires that members of the scientific community register for access to the repository.
URL: https://www.cos.io/products/osf-registries?hsCtaTracking=6f4c9f67-31b7-477a-a8b4-2fbe385ff3fe%7C21b2d2be-373c-4d61-9210-da8fbc1f2962